CLINICAL TRIAL: NCT02496715
Title: Randomized, Parallel, Placebo-controlled, Multiple Dose, Multicenter Study to Compare the Efficacy of Fluticasone/Salmeterol (Test) to Advair® Diskus (GSK) in Adult Asthma Patients
Brief Title: Randomized, Placebo-controlled Study Comparing Efficacy of Fluticasone/Salmeterol Combination to Advair in Asthmatics
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Development terminated.
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT-2014-075
Record Dates: First submitted 2015-07-01; First posted 2015-07-14 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1 (Experimental): Generic fluticasone propionate 100 mcg / salmeterol 50 mcg. Single puff, twice daily (approximately every 12 hr) for 4 weeks
  Interventions: Drug: Generic fluticasone propionate 100 mcg / salmeterol 50 mcg
- Treatment 2 (Experimental): Advair 100/50 Diskus pMDI containing fluticasone propionate 100mcg / salmeterol 50 mcg. Single puff, twice daily (approximately every 12 hr) for 4 weeks
  Interventions: Drug: Fluticasone propionate 100 mcg / salmeterol 50 mcg
- Treatment 3 (Placebo Comparator): Placebo inhalation. Single puff, twice daily (approximately every 12 hr) for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate 100 mcg / salmeterol 50 mcg — Brand inhaler containing pMDI containing fluticasone and salmeterol
  Other Names: Advair
  Arms: Treatment 2
Drug: Generic fluticasone propionate 100 mcg / salmeterol 50 mcg — Generic inhaler containing pMDI containing fluticasone and salmeterol
  Other Names: Generic Test
  Arms: Treatment 1
Drug: Placebo — Placebo inhaler
  Arms: Treatment 3

SUMMARY:
This is a pivotal trial that will examine therapeutic equivalence (BE) of a new generic fixed-dose combination product containing fluticasone propionate 100 mcg / salmeterol 50 mcg (as xinafoate salt) and reference listed drug (RLD) Advair® Diskus 100/50 in adult patients with chronic but stable asthma as defined in the National Asthma Education and Prevention Program Expert Panel Report 3 (NAEPP 3) guidelines

DETAILED DESCRIPTION:
This pivotal trial will examine therapeutic equivalence of a new generic fixed-dose combination product containing fluticasone propionate 100 mcg / salmeterol 50 mcg (as xinafoate salt) and reference listed drug (RLD) Advair® Diskus 100/50 in adult patients with chronic but stable asthma as defined in National Asthma Education and Prevention Program Expert Panel Report 3 (NAEPP 3) guidelines [2]. To ensure adequate study sensitivity the test and reference products should both be statistically superior to placebo (p<0.05) with regard to the BE study primary endpoints.

A secondary study objective is the safety and tolerability of the test compound.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects of non-childbearing or of childbearing potential committed to consistent and correct use of an acceptable method of birth control
* Diagnosed with asthma, as defined by the National Asthma Education and Prevention Program (NAEPP),5 at least 6 months prior to screening
* Moderate-to-severe asthma with a pre-bronchodilator FEV1 of >45% and <85% of predicted normal, measured at least 6 hours after short-acting β agonist (SABA)and at least 24 hours after the last dose of long-acting β agonist (LABA), at the screening visit and on the day of treatment
* >15% and >0.20 L reversibility of FEV1 within 30 minutes following 360 mcg of albuterol inhalation (pMDI)
* Patients should be stable on their chronic asthma treatment regimen for at least 4 weeks prior to enrollment
* Currently non-smoking; having not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and having < 10 pack-years of historical use
* Able to replace current regularly scheduled short-acting β agonists (SABAs) with salbutamol/albuterol inhaler for use only on an as-needed basis for the duration of the study (subjects should be able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits)
* Willing to discontinue their asthma medications (inhaled corticosteroids and long-acting β agonists) during the run-in period and for the remainder of the study
* Willingness to give their written informed consent to participate in the study

Exclusion Criteria:

* Life-threatening asthma, defined as a history of asthma episodes(s) requiring intubation, and/or associated with hypercapnia, respiratory arrest or hypoxic seizures, asthma-related syncopal episodes(s), or hospitalizations within the past year or during the run-in period
* Significant respiratory disease other than asthma (chronic obstructive pulmonary disease (COPD), interstitial lung disease, etc.)
* Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition,historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that, in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study
* Patients who required systemic corticosteroids (for any reason) within the past 4 weeks
* Hypersensitivity to any sympathomimetic drug (e.g., formoterol or albuterol) or any inhaled, intranasal, or systemic corticosteroid therapy
* Patients currently receiving β-blockers

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Baseline-corrected area under the serial Forced Expiratory Volume in the first second (FEV1)-time effect curve calculated from time zero to 12 hours on the first day of the treatment | up to 12 hours
  Baseline-corrected area under the serial FEV1-time effect curve calculated from time zero to 12 hours on the first day of the treatment (Visit 2, Day 1) to assess equivalence of test drug with reference listed drug (RLD) Advair® Diskus® 100/50, and to assess superiority over placebo

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) results at the times of FEV1 measurements | Day 1 and Day 28
Daily rescue medication used | 8 weeks
  The type and frequency of rescue medication used
Number and type of adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Beverley Patterson, PhD, Study Director — Actavis Inc.